CLINICAL TRIAL: NCT04658394
Title: Effect of Individual Reminiscence Therapy in the Elderly People With Neurocognitive Disorders: A Multicentre Randomised Controlled Trial in Azores Archipelago
Brief Title: Effect of Individual Reminiscence Therapy in the Elderly People With Neurocognitive Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rsocialform - Geriatria, Lda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21112020
Record Dates: First submitted 2020-11-24; First posted 2020-12-08 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-01

CONDITIONS: Dementia; Neurocognitive Disorders; Cognitive Impairment; Cognitive Dysfunction; Cognitive Decline
Keywords: older adults; dementia; reminiscence therapy; quality of life; cognition; neurocognitive disorders; individual therapy; non-pharmacological therapy; randomised controlled trial; mood; depression; anxiety; memory
MeSH Terms: conditions — Dementia; Neurocognitive Disorders; Cognitive Dysfunction; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants who meet the inclusion criteria will be randomly assigned to the intervention group receiving RT or to a control group receiving treatment as usual. Participants in the intervention group will participate in two RT sessions per week for 13 weeks besides their treatment as usual. The sessions will be based on the Book of the Past and the Present and they will follow the same protocol in every participant institution.
  Interventions: Other: Reminiscence therapy
- Control Group (No Intervention): Participants assigned to the control group will maintain their usual treatment in the institution, participating in the activities previously assigned to their individual care plan.

INTERVENTIONS:
Other: Reminiscence therapy — Intervention group will receive two RT sessions per week for 13 weeks. RT sessions will last approximately 50 minutes and will be developed according to the following structure: · Welcome to the patient and reality orientation therapy (7 minutes) · Conducting the main activity of reminiscence (40 minutes) · Closure, thank you for the participation and farewell until the next session (3 minutes) Reminiscence therapy sessions will have an individual format and will be conducted by a therapist previously trained in the protocol and the principles of RT. The Reminiscence activities of each session will be carried out following the protocol proposed in the Book of the Past and the Present.
  Arms: Intervention Group

SUMMARY:
This research aims to evaluate the ability of individual reminiscence therapy (RT), using a simple reminiscence format, to improve the overall cognitive function, memory, emotional status and quality of life (QoL) of older adults with neurocognitive disorders (NCD) attending social care and support services. A multicentre randomised controlled trial (RCT) is proposed in Azores archipelago with repeated measures (pre-intervention, post-intervention and follow-up). Intervention group will hold 26 individual RT sessions, twice a week for 13 weeks. Control group participants will maintain their treatment as usual. Make a subsample analysis of the main clinical diagnoses, and compare the results of sample and subsample with a previous study that had the same intervention protocol.

DETAILED DESCRIPTION:
Neurocognitive disorder (NCD) is one of the main causes of disability among older adults and its prevalence is increasing due to the ageing of the population. It is estimated that globally, neurocognitive disorders affect 44.35 million people and it is expected that by the year 2050 the number of those affected worldwide will triple up to 135.46 million.

The absence of an effective pharmacological treatment that halts or delays the development of the disease has aroused interest in non-pharmacological therapies (NPT) as a complement to pharmacological treatment that can improve the quality of life of people with neurocognitive disorders. One of the most researched NPT and with the greatest tradition in this field is Reminiscence Therapy (RT).

RT implies the discussion of past activities, events and experiences, usually with the help of triggers (e.g., photographs, home objects and other familiar items from the past, music, any object or stimulus) that serve to stimulate memories. In its application to dementias, RT is based on the fact that the memory deficit of people with dementia implies that they are able to remember events from their past life, especially from childhood to early adulthood, but not newer facts. It focuses on preserved capacities and memories, promotes communication and enables the person to connect with his past and recover his sense of personal identity. In this way, the RT can be understood as an intervention on the edge of those of cognitive orientation and those centred on emotion, with potential interactive effects on autobiographical memory and psychological well-being.

In simplified form, there are at least two approaches to RT. The first approach as a "life review" where participants are guided through significant experiences of their biography trying to give meaning to their lives. This type of RT is more structured and is usually conducted in an individual format. It may involve the production of "life books". This approach is considered to have an integrative function aimed at achieving a sense of validation, coherence and reconciliation with one's past. Another approach that call general or simple reminiscence, implies the stimulation of autobiographical memory during conversations on specific themes of the past (e.g, holidays, food and drink, work) using stimulus to trigger memories. It has been described as an unstructured autobiographical memory narration. This reminiscence format can be conducted both individually and in groups and promotes communication between participants who share their memories and stories.

In either format that RT is applied on, the introduction of triggering stimulus (e.g., photographs, music, old objects) to help memory is considered fundamental. These triggers can be generic, reflecting common experiences in the lives of people relevant to their age group (e.g., a school manual can serve as a reminder of the experience during their school stage), or specific, with stimulus related to the person's own experiences (e.g., photographs of an important vital event such as their wedding day or a journey during their youth).

As for the effectiveness of RT, according to a recent review by Cochrane, there is some evidence on its positive effects on cognition, QoL, communication and possibly on the mood of people with dementia, even if the benefits are small. Despite the distinction between the two different approaches to RT (general reminiscence vs. life history), the therapy modality does not seem to be as important to achieve positive effects as the individual or group format of the sessions and the context in which the intervention is administered (people living in the community or institutionalised).

In particular, according to the results of the review study, the RT seems to be able to generate a small benefit on cognitive function immediately after the intervention, although it usually does not continue after a longer follow-up period. Regarding the administration format, the individual RT seems slightly superior in its effects on cognition both immediately and after a follow-up period. In any case, its effects seem comparable to those of other cognitive stimulation modalities.

As for the effect of RT on quality of life (QoL), an individual RT study based on life review, showed an improvement in Qol-AD. The effects with a group modality do not seem consistent, showing little or no effect on QoL, although the key factor may be the context of application (community vs. institution), with better group RT results in institutionalised patients.

In a multicentre study conducted in Portugal with older adults with neurocognitive disorders, in individual format, there was a significant effect on the overall cognition, memory and QoL of the participants.

Group RT was associated with a likely effect on communication both after the intervention and in the follow-up. This effect was not replicated in the individual RT, with uncertain results.

Finally, despite the evidence on the effect of RT on the mood of elderly people without dementia, in the case of people with dementia only a small effect on mood was found for those participating in individual RT. In the portuguese multicentre studies there were no significant differences in depressive symptomatology.

Based on the above, this research proposal aims to evaluate the ability of individual RT within a general reminiscence format, to improve overall cognitive function, in particular memory, emotional state (depression and anxiety) and QoL of older adults with neurocognitive disorders attending social care and support services in the Azores archipelago.

It is proposed to evaluate the efficacy of the intervention in the endpoint assessment and the duration of the effects at three months follow-up. Furthermore, an analysis of results based on the diagnosis of the participants is proposed for those diagnoses with sufficient representation in the sample (more than 20 cases in each group). Additionally, it is proposed to analyze the factors that predict the response to the intervention (responder analysis). Finally, the results of this study will be compared and can be analyzed together with those of a previous study that used the same individual RT program and the same experimental design (clinicaltrials.gov ID: NCT04047238).

ELIGIBILITY:
Inclusion Criteria:

* Having a formal diagnosis of a neurocognitive disorder according to Diagnostic and Statistical Manual of Mental Disorders, fifth edition [DSM-5] criteria (participants diagnosis will be confirm in their health records at the institution).
* Having delivered the informed consent form, duly completed and signed, after prior information.
* Being able to communicate and understand.
* Possibility of gathering information about the participant's life history through family members or usual caregivers, using the socio-family questionnaire designed for that purpose.
* Being 65 years of age or older.
* Being a native Portuguese speaker.
* Regularly attending an institution that provides social care and support services for older adults (including people living in long-term care centres, people attending day and social centres and people receiving home support services).

Exclusion Criteria:

* Suffering from an acute or severe illness that prevent participation in the intervention sessions.
* Severe sensory and physical limitations that prevent participation.
* Low level of consciousness and minimal attention span.
* Presence of severe neuropsychiatric symptoms, such as agitation, psychosis, severe depressive and anxiety symptoms, apathy, or presence of uncontrolled delirium that prevent participation in the sessions.
* Traumatic life history or marked by adverse events that discourage participation in RT sessions; history of adverse reactions during RT sessions or similar activities.
* Have a serious or total functional dependence (assessed through the Barthel index).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Cognitive functioning evaluated through Mini-Mental State Examination [MMSE] | baseline
  Cognitive functioning is assessed using the MMSE which is a gold standard for assessing global cognitive function. Scores range from 0 to 30, with higher scores indicating better cognitive functioning.
Change in cognitive functioning evaluated through Mini-Mental State Examination [MMSE] | 13 weeks after the beginning of the intervention
  Cognitive functioning is assessed using the MMSE which is a gold standard for assessing global cognitive function. Scores range from 0 to 30, with higher scores indicating better cognitive functioning.
Change in cognitive functioning evaluated through Mini-Mental State Examination [MMSE] | 12 weeks after end of intervention
  Cognitive functioning is assessed using the MMSE which is a gold standard for assessing global cognitive function. Scores range from 0 to 30, with higher scores indicating better cognitive functioning.

SECONDARY OUTCOMES:
Quality of life evaluated through Quality of Life - Alzheimer's Disease [QoL-AD] | baseline
  The QoL-AD is used to assess quality of life. This 13-item scale assesses the quality of life in people diagnosed with dementia, gathering information from the patient about the following domains: perceived health, mood, physical condition, interpersonal relationships, hobbies, decision-making skills, and life as a whole. Scores range from 13 to 52, with higher scores indicating better quality of life. It has good psychometric characteristics and its use has been recommended to evaluate psychosocial interventions.
Change in quality of life evaluated through Quality of Life - Alzheimer's Disease [QoL-AD] | 13 weeks after the beginning of the intervention
  The QoL-AD is used to assess quality of life. This 13-item scale assesses the quality of life in people diagnosed with dementia, gathering information from the patient about the following domains: perceived health, mood, physical condition, interpersonal relationships, hobbies, decision-making skills, and life as a whole. Scores range from 13 to 52, with higher scores indicating better quality of life. It has good psychometric characteristics and its use has been recommended to evaluate psychosocial interventions.
Change in quality of life evaluated through Quality of Life - Alzheimer's Disease [QoL-AD] | 12 weeks after end of intervention
  The QoL-AD is used to assess quality of life. This 13-item scale assesses the quality of life in people diagnosed with dementia, gathering information from the patient about the following domains: perceived health, mood, physical condition, interpersonal relationships, hobbies, decision-making skills, and life as a whole. Scores range from 13 to 52, with higher scores indicating better quality of life. It has good psychometric characteristics and its use has been recommended to evaluate psychosocial interventions.
Anxiety symptomatology assessed through the Geriatric Anxiety Inventory [GAI] | baseline
  It assesses, in several contexts, the severity of anxiety symptoms in the older adults. It consists in 20 dichotomous response items (I agree/disagree) and refers to the subject's feelings in the week prior to the evaluation. One (1) point is assigned to each agree answer and the overall score is obtained by adding the scores of all items. Scores over 10/11 points indicate symptoms of severe anxiety.
Change in anxiety symptomatology assessed through the Geriatric Anxiety Inventory [GAI] | 13 weeks after the beginning of the intervention
  It assesses, in several contexts, the severity of anxiety symptoms in the older adults. It consists in 20 dichotomous response items (I agree/disagree) and refers to the subject's feelings in the week prior to the evaluation. One (1) point is assigned to each agree answer and the overall score is obtained by adding the scores of all items. Scores over 10/11 points indicate symptoms of severe anxiety.
Change in anxiety symptomatology assessed through the Geriatric Anxiety Inventory [GAI] | 12 weeks after end of intervention
  It assesses, in several contexts, the severity of anxiety symptoms in the older adults. It consists in 20 dichotomous response items (I agree/disagree) and refers to the subject's feelings in the week prior to the evaluation. One (1) point is assigned to each agree answer and the overall score is obtained by adding the scores of all items. Scores over 10/11 points indicate symptoms of severe anxiety.
Mood assessed through the Geriatric Depression Scale-15 [GDS-15] | baseline
  The GDS-15 is used to measure mood. It is considered a reliable tool to screen depressive symptoms in older people. With a dichotomous format (yes/no answers), this scale assesses depression in older people. Scores range from 0 to 15, with higher scores indicating more severe depressive symptoms.
Change in mood assessed through the Geriatric Depression Scale-15 [GDS-15] | 13 weeks after the beginning of the intervention
  The GDS-15 is used to measure mood. It is considered a reliable tool to screen depressive symptoms in older people. With a dichotomous format (yes/no answers), this scale assesses depression in older people. Scores range from 0 to 15, with higher scores indicating more severe depressive symptoms.
Change in mood assessed through the Geriatric Depression Scale-15 [GDS-15] | 12 weeks after end of intervention
  The GDS-15 is used to measure mood. It is considered a reliable tool to screen depressive symptoms in older people. With a dichotomous format (yes/no answers), this scale assesses depression in older people. Scores range from 0 to 15, with higher scores indicating more severe depressive symptoms.
Executive functions evaluated throught Frontal Assessment Battery [FAB] | baseline
  The FAB is used to assess executive function in several subtests: conceptualization, mental flexibility, motor programming, sensitivity to interference, inhibitory control, and environmental autonomy. Scores range from 0 to 18, with higher scores indicating better executive functioning.
Change in executive functions evaluated throught Frontal Assessment Battery [FAB] | 13 weeks after the beginning of the intervention
  The FAB is used to assess executive function in several subtests: conceptualization, mental flexibility, motor programming, sensitivity to interference, inhibitory control, and environmental autonomy. Scores range from 0 to 18, with higher scores indicating better executive functioning.
Change in executive functions evaluated throught Frontal Assessment Battery [FAB] | 12 weeks after end of intervention
  The FAB is used to assess executive function in several subtests: conceptualization, mental flexibility, motor programming, sensitivity to interference, inhibitory control, and environmental autonomy. Scores range from 0 to 18, with higher scores indicating better executive functioning.
Memory function evaluated through Memory Alteration Test [MAT] | baseline
  The MAT is used to assess memory function. It is an easy and quick instrument that assesses five memory domains: temporal orientation, encoding, semantic memory, free recall, and cued recall. Total scores range from 0 to 50, with higher scores indicating better memory. It has good psychometric properties and is highly sensitive to mild cognitive decline.
Change in memory function evaluated through Memory Alteration Test [MAT] | 13 weeks after the beginning of the intervention
  The MAT is used to assess memory function. It is an easy and quick instrument that assesses five memory domains: temporal orientation, encoding, semantic memory, free recall, and cued recall. Total scores range from 0 to 50, with higher scores indicating better memory. It has good psychometric properties and is highly sensitive to mild cognitive decline.
Change in memory function evaluated through Memory Alteration Test [MAT] | 12 weeks after end of intervention
  The MAT is used to assess memory function. It is an easy and quick instrument that assesses five memory domains: temporal orientation, encoding, semantic memory, free recall, and cued recall. Total scores range from 0 to 50, with higher scores indicating better memory. It has good psychometric properties and is highly sensitive to mild cognitive decline.

OTHER OUTCOMES:
Sociodemographic information gathered through the sociodemographic questionnaire | baseline
  Participants' answers in the sociodemographic questionnaire designed specifically for this study. It gathers information about gender, age, marital status, formal education, which social response the participant attends, medical comorbidities and cognitive symptoms and will be administered to all participants.
Functional dependence evaluated through Barthel Index [IB] | before baseline (exclusion criteria)
  This is a 10-item self-administered scale that evaluates the functional capacity to conduct daily life activities. The activities are quoted differently, 0, 1, 2 or 3 points can be assigned. The total score ranges from 0 (totally dependent) to 20 (totally independent), with a total of 0-8 being total dependency; 9-12 being serious dependency; 13-19 being moderate dependency; 20 being total independence. This instrument has item-total correlations between .66 and .93, and has a high internal consistency (Cronbach alpha of .96).

CONTACTS AND LOCATIONS:
Overall Officials: Susana I Justo Henriques, PhD, Principal Investigator — Nursing School of Coimbra; Enrique Pérez Sáez, PhD, Principal Investigator — National Reference Centre for Alzheimer's and Dementia Care, Imserso, Spain; João L. Alves Apóstolo, PhD, Principal Investigator — Nursing School of Coimbra
Locations (13):
- Portugal (13):
  - Rsocialform - Geriatria, Lda., Mealhada, Aveiro District
  - Santa Casa da Misericórdia da Horta, Horta, Faial
  - Santa Casa da Misericórdia de Santa Cruz das Flores, Santa Cruz das Flores, Flores
  - Santa Casa da Misericórdia de Lajes do Pico, Lajes, Pico
  - Santa Casa da Misericórdia da Madalena do Pico, Madalena, Pico
  - Santa Casa da Misericórdia de Vila do Porto, Vila do Porto, Santa Maria
  - Santa Casa da Misericórdia da Calheta, Calheta, São Jorge
  - Casa de Repouso João Inácio de Sousa, Velas, São Jorge
  - Casa do Povo de Arrifes, Arrifes, São Miguel
  - Casa do Povo da Maia, Maia, São Miguel
  - Lar Luis Soares de Sousa de Ponta Delgada, Ponta Delgada, São Miguel
  - Santa Casa da Misericórdia de Angra do Heroísmo, Angra do Heroísmo, Terceira
  - Lar D. Pedro V, Praia da Vitória, Terceira

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akanuma K, Meguro K, Meguro M, Sasaki E, Chiba K, Ishii H, Tanaka N. Improved social interaction and increased anterior cingulate metabolism after group reminiscence with reality orientation approach for vascular dementia. Psychiatry Res. 2011 Jun 30;192(3):183-7. doi: 10.1016/j.pscychresns.2010.11.012. Epub 2011 May 4. PMID 21543189
- [Background] Amieva H, Robert PH, Grandoulier AS, Meillon C, De Rotrou J, Andrieu S, Berr C, Desgranges B, Dubois B, Girtanner C, Joel ME, Lavallart B, Nourhashemi F, Pasquier F, Rainfray M, Touchon J, Chene G, Dartigues JF. Group and individual cognitive therapies in Alzheimer's disease: the ETNA3 randomized trial. Int Psychogeriatr. 2016 May;28(5):707-17. doi: 10.1017/S1041610215001830. Epub 2015 Nov 17. PMID 26572551
- [Background] Apóstolo JLA, Bobrowicz-Campos EM, dos Reis IAC, Henriques SJ, Correia CAV. Exploring the screening capacity of the European Portuguese version of the 15-item Geriatric Depression Scale. Revista de Psicopatología y Psicología Clínica. 2018; 23: 99-107. doi: 10.5944/rppc.vol.23.num.2.2018.21050
- [Background] Apóstolo J, Loureiro L, Reis I, Silva I, Cardoso D, Sfetcu R. Contribution to the adaptation of the Geriatric Depression Scale -15 into Portuguese. Revista de Enfermagem Referência. 2014; IV(3): 65-73. doi: 10.12707/RIV14033
- [Background] Araújo F, Pais-Ribeiro J, Oliveira A, Pinto C. Validação do índice de Barthel numa amostra de idosos não institucionalizados. Revista Portuguesa de Saúde Pública. 2007; 25(2): 59-66.
- [Background] Serrani Azcurra DJ. A reminiscence program intervention to improve the quality of life of long-term care residents with Alzheimer's disease: a randomized controlled trial. Braz J Psychiatry. 2012 Dec;34(4):422-33. doi: 10.1016/j.rbp.2012.05.008. PMID 23429813
- [Background] Barrios H, Verdelho A, Narciso S, Goncalves-Pereira M, Logsdon R, de Mendonca A. Quality of life in patients with cognitive impairment: validation of the Quality of Life-Alzheimer's Disease scale in Portugal. Int Psychogeriatr. 2013 Jul;25(7):1085-96. doi: 10.1017/S1041610213000379. Epub 2013 Mar 27. PMID 23534370
- [Background] Caddell LS, Clare L. The impact of dementia on self and identity: a systematic review. Clin Psychol Rev. 2010 Feb;30(1):113-26. doi: 10.1016/j.cpr.2009.10.003. PMID 19896760
- [Background] Charlesworth G, Burnell K, Crellin N, Hoare Z, Hoe J, Knapp M, Russell I, Wenborn J, Woods B, Orrell M. Peer support and reminiscence therapy for people with dementia and their family carers: a factorial pragmatic randomised trial. J Neurol Neurosurg Psychiatry. 2016 Nov;87(11):1218-1228. doi: 10.1136/jnnp-2016-313736. Epub 2016 Aug 12. PMID 27521377
- [Background] Dempsey L, Murphy K, Cooney A, Casey D, O'Shea E, Devane D, Jordan F, Hunter A. Reminiscence in dementia: a concept analysis. Dementia (London). 2014 Mar 1;13(2):176-92. doi: 10.1177/1471301212456277. Epub 2012 Aug 17. PMID 24599812
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Freitas S, Simoes MR, Alves L, Santana I. The Relevance of Sociodemographic and Health Variables on MMSE Normative Data. Appl Neuropsychol Adult. 2015;22(4):311-9. doi: 10.1080/23279095.2014.926455. Epub 2014 Dec 22. PMID 25531579
- [Background] Gonzalez J, Mayordomo T, Torres M, Sales A, Melendez JC. Reminiscence and dementia: a therapeutic intervention. Int Psychogeriatr. 2015 Oct;27(10):1731-7. doi: 10.1017/S1041610215000344. Epub 2015 Mar 13. PMID 25765779
- [Background] Guerreiro M, Silva AP, Botelho MA, Leitão O, Castro-Caldas A, Garcia C. Adaptação à população portuguesa da tradução do Mini Mental State Examination (MMSE). Revista Portuguesa de Neurologia. 1994; 1: 9-10.
- [Background] Haight BK, Gibson F, Michel Y. The Northern Ireland life review/life storybook project for people with dementia. Alzheimers Dement. 2006 Jan;2(1):56-8. doi: 10.1016/j.jalz.2005.12.003. PMID 19595856
- [Background] Henriques SIJ. Livro do Passado e do Presente [Book of the Past and the Present]. Mealhada, Replicar Socialform; 2018.
- [Background] Justo-Henriques SI, Perez-Saez E, Alves Apostolo JL. Multicentre randomised controlled trial about the effect of individual reminiscence therapy in older adults with neurocognitive disorders. Int J Geriatr Psychiatry. 2021 May;36(5):704-712. doi: 10.1002/gps.5469. Epub 2020 Nov 17. PMID 33176394
- [Background] Justo-Henriques SI, Pérez-Sáez E, Apóstolo JLA. Individual intervention protocol based on reminiscence therapy for older people with neurocognitive disorders. Revista de Enfermagem de Referência. 2020; 5(3): e20043. doi: 10.12707/RV20043
- [Background] Kirk M, Berntsen D. A short cut to the past: Cueing via concrete objects improves autobiographical memory retrieval in Alzheimer's disease patients. Neuropsychologia. 2018 Feb;110:113-122. doi: 10.1016/j.neuropsychologia.2017.06.034. Epub 2017 Jul 1. PMID 28676268
- [Background] Kirk M, Rasmussen KW, Overgaard SB, Berntsen D. Five weeks of immersive reminiscence therapy improves autobiographical memory in Alzheimer's disease. Memory. 2019 Apr;27(4):441-454. doi: 10.1080/09658211.2018.1515960. Epub 2018 Sep 8. PMID 30198380
- [Background] Lai CK, Chi I, Kayser-Jones J. A randomized controlled trial of a specific reminiscence approach to promote the well-being of nursing home residents with dementia. Int Psychogeriatr. 2004 Mar;16(1):33-49. doi: 10.1017/s1041610204000055. PMID 15190995
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Quality of life in Alzheimer's disease: Patient and caregiver reports. Journal of Mental Health and Aging. 1999; 5: 21-32.
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] Moniz-Cook E, Vernooij-Dassen M, Woods R, Verhey F, Chattat R, De Vugt M, Mountain G, O'Connell M, Harrison J, Vasse E, Droes RM, Orrell M; INTERDEM group. A European consensus on outcome measures for psychosocial intervention research in dementia care. Aging Ment Health. 2008 Jan;12(1):14-29. doi: 10.1080/13607860801919850. PMID 18297476
- [Background] Morgado J, Rocha CS, Maruta C, Guerreiro M, Martins IP. Novos valores normativos do Mini-Mental State Examination. Sinapse. 2009; 2: 10-16.
- [Background] O'Shea E, Devane D, Cooney A, Casey D, Jordan F, Hunter A, Murphy E, Newell J, Connolly S, Murphy K. The impact of reminiscence on the quality of life of residents with dementia in long-stay care. Int J Geriatr Psychiatry. 2014 Oct;29(10):1062-70. doi: 10.1002/gps.4099. Epub 2014 Mar 14. PMID 24633858
- [Background] Pachana NA, Byrne GJ, Siddle H, Koloski N, Harley E, Arnold E. Development and validation of the Geriatric Anxiety Inventory. Int Psychogeriatr. 2007 Feb;19(1):103-14. doi: 10.1017/S1041610206003504. PMID 16805925
- [Background] Pinquart M, Duberstein PR, Lyness JM. Effects of psychotherapy and other behavioral interventions on clinically depressed older adults: a meta-analysis. Aging Ment Health. 2007 Nov;11(6):645-57. doi: 10.1080/13607860701529635. PMID 18074252
- [Background] Prince M, Guerchet M, Prina M. World Alzheimer Report 2015. The global impact of dementia: An analysis of prevalence, incidence, cost and trends. London: Alzheimer´s Disease International (ADI); 2015. http://www.worldalzreport2015.org/downloads/world-alzheimer-report-2015.pdf
- [Background] Rami L, Molinuevo JL, Sanchez-Valle R, Bosch B, Villar A. Screening for amnestic mild cognitive impairment and early Alzheimer's disease with M@T (Memory Alteration Test) in the primary care population. Int J Geriatr Psychiatry. 2007 Apr;22(4):294-304. doi: 10.1002/gps.1672. PMID 16998781
- [Background] Ribeiro O, Paul C, Simoes MR, Firmino H. Portuguese version of the Geriatric Anxiety Inventory: transcultural adaptation and psychometric validation. Aging Ment Health. 2011 Aug;15(6):742-8. doi: 10.1080/13607863.2011.562177. Epub 2011 Jun 9. PMID 21656405
- [Background] Sarkamo T, Tervaniemi M, Laitinen S, Numminen A, Kurki M, Johnson JK, Rantanen P. Cognitive, emotional, and social benefits of regular musical activities in early dementia: randomized controlled study. Gerontologist. 2014 Aug;54(4):634-50. doi: 10.1093/geront/gnt100. Epub 2013 Sep 5. PMID 24009169
- [Background] Subramaniam P, Woods B. Towards the therapeutic use of information and communication technology in reminiscence work for people with dementia: a systematic review. International Journal of Computers in Healthcare. 2010; 1: 106-125. doi: 10.1504/IJCIH.2010.037457.
- [Background] Subramaniam P, Woods B. The impact of individual reminiscence therapy for people with dementia: systematic review. Expert Rev Neurother. 2012 May;12(5):545-55. doi: 10.1586/ern.12.35. PMID 22550983
- [Background] Subramaniam P, Woods B, Whitaker C. Life review and life story books for people with mild to moderate dementia: a randomised controlled trial. Aging Ment Health. 2014;18(3):363-75. doi: 10.1080/13607863.2013.837144. Epub 2013 Sep 24. PMID 24063317
- [Background] Tadaka E, Kanagawa K. Effects of reminiscence group in elderly people with Alzheimer disease and vascular dementia in a community setting. Geriatrics & Gerontology International. 2007; 7: 167-173. doi: 10.1111/j.1447-0594.2007.00381.x
- [Background] Thorgrimsen L, Schweitzer P, Orrell M. Evaluating reminiscence for people with dementia: A pilot study. The Arts in Psychotherapy. 2002; 29: 93-97. doi: 10.1016/S0197-4556(01)00135-6
- [Background] Westerhof GJ, Bohlmeijer E, Webster JD. Reminiscence and mental health: A review of recent progress in theory, research and interventions. Ageing & Society. 2010; 30: 697-721. doi: 10.1017/S0144686X09990328
- [Background] Wong PT, Watt LM. What types of reminiscence are associated with successful aging? Psychol Aging. 1991 Jun;6(2):272-9. doi: 10.1037//0882-7974.6.2.272. PMID 1863396
- [Background] Woods B, O'Philbin L, Farrell EM, Spector AE, Orrell M. Reminiscence therapy for dementia. Cochrane Database Syst Rev. 2018 Mar 1;3(3):CD001120. doi: 10.1002/14651858.CD001120.pub3. PMID 29493789
- [Background] Woods B, Spector A, Jones C, Orrell M, Davies S. Reminiscence therapy for dementia. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD001120. doi: 10.1002/14651858.CD001120.pub2. PMID 15846613
- [Background] Woods RT, Bruce E, Edwards RT, Elvish R, Hoare Z, Hounsome B, Keady J, Moniz-Cook ED, Orgeta V, Orrell M, Rees J, Russell IT. REMCARE: reminiscence groups for people with dementia and their family caregivers - effectiveness and cost-effectiveness pragmatic multicentre randomised trial. Health Technol Assess. 2012;16(48):v-xv, 1-116. doi: 10.3310/hta16480. PMID 23211271
- [Background] Woods RT, Bruce E, Edwards RT, Hounsome B, Keady J, Moniz-Cook ED, Orrell M, Russell IT. Reminiscence groups for people with dementia and their family carers: pragmatic eight-centre randomised trial of joint reminiscence and maintenance versus usual treatment: a protocol. Trials. 2009 Jul 30;10:64. doi: 10.1186/1745-6215-10-64. PMID 19642992
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Lima CF, Meireles LP, Fonseca R, Castro SL, Garrett C. The Frontal Assessment Battery (FAB) in Parkinson's disease and correlations with formal measures of executive functioning. J Neurol. 2008 Nov;255(11):1756-61. doi: 10.1007/s00415-008-0024-6. Epub 2008 Sep 25. PMID 18821046
- [Background] Dubois B, Slachevsky A, Litvan I, Pillon B. The FAB: a Frontal Assessment Battery at bedside. Neurology. 2000 Dec 12;55(11):1621-6. doi: 10.1212/wnl.55.11.1621. PMID 11113214
- [Background] Perez-Saez E, Justo-Henriques SI, Alves Apostolo JL. Multicenter randomized controlled trial of the effects of individual reminiscence therapy on cognition, depression and quality of life: Analysis of a sample of older adults with Alzheimer's disease and vascular dementia. Clin Neuropsychol. 2022 Oct;36(7):1975-1996. doi: 10.1080/13854046.2021.1871962. Epub 2021 Jan 19. PMID 33467972